CLINICAL TRIAL: NCT02917356
Title: The Effect of Laying on of Hands on the Pain, Joint Stiffness and Functional Capacity of Older Women With Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: The Effect of "Laying on of Hands" in Older Women With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Principal Investigator, Giancarlo Lucchetti, MD, PhD, Federal University of Juiz de Fora
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE52623115.0.0000.5147
Record Dates: First submitted 2016-09-25; First posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Knee Osteoarthritis
Keywords: Healing touch; Faith Healing; Pain; Joint stiffness; Functional status; Mental health; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Psychological Well-Being; Osteoarthritis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Spiritual laying on of hands group (Experimental): * Spiritist Passe - performed by spiritual healers from the religion Spiritism (5 min, once a week, for 8 weeks)
  * Physical therapy: Kinesiotherapy (45 min, twice a week, for 8 weeks)
  Interventions: Other: Spiritual laying on of hands (SP)
- Non-spiritual Laying on of Hands group (Active Comparator): * Non-spiritual Laying on of Hands - performed by lay persons (5 min, once a week, for 8 weeks)
  * Physical therapy: Kinesiotherapy (45 min, twice a week, for 8 weeks)
  Interventions: Other: Non-spiritual Laying on of Hands
- Control Group (CG) (Sham Comparator): * Sham/ Control Group (CG) - performed by lay persons. They will stay in the room and move slowly and randomly in order to sham the presence of someone performing the laying on of hands. However, they will not perform the laying on of hands (5 min, once a week, for 8 weeks)
  * Physical therapy: Kinesiotherapy (45 min, twice a week, for 8 weeks)
  Interventions: Other: Control group

INTERVENTIONS:
Other: Spiritual laying on of hands (SP) — The SP will be applied after physical therapy (kinesiotherapy). Spiritual healers from Spiritism will perform the SP. In order to produce a culturally acceptable environment, the Spiritist therapists will 'prepare' the environment by praying for 5 minutes. The Spiritist therapists will hold both hands 10-15 cm above the patients' head. Then, they will longitudinally lower their hands starting from the patients' head towards their legs, for four times. Subsequently, the therapists shall lay their hands on patients' head and on their knees. The therapists will remain silent during these procedures and try to 'heal' the patients. The subjects will remain in a seated position, blindfolded with dark-blinded goggles, and will receive the following verbal command: "Relax and calm your mind."
  Other Names: Spiritist Healing; Spiritist passe
  Arms: Spiritual laying on of hands group
Other: Non-spiritual Laying on of Hands — The non-spiritual laying on of hands will be applied after physical therapy (kinesiotherapy), for 5 minutes, without touching the patients and without 'preparing' the environment. They will hold their hands 10-15 cm above patient's head and will focus on healing the patients. They will visualize the following sentence: "I want you to heal"; without saying prayers or invocations. The subjects will remain in a seated position, blindfolded with dark-blinded goggles, and will receive the following verbal command: "Relax and calm your mind."
  Arms: Non-spiritual Laying on of Hands group
Other: Control group — The patients will be subjected to physical therapy (kinesiotherapy), only. However, they will be accompanied by people who will stay in the room and move slowly and randomly in order to sham the presence of someone performing the laying on of hands. However, they will not perform the laying on of hands. These people will not focus on healing the patients and they will be asked to mentally count 5 minutes while they are with the patients. The subjects will remain in a seated position, blindfolded with dark-blinded goggles, and will receive the following verbal command: "Relax and calm your mind."
  Arms: Control Group (CG)

SUMMARY:
Osteoarthritis (OA) is the most common form of chronic degenerative joint disease, as well as the main cause of pain and disability in older persons worldwide. The limited results of physical therapy in OA makes OA patients potential candidates for complementary therapies, such as laying on of hands. The present study aims to investigate the effect of Laying on of Hands on the Pain, Joint Stiffness and Functional Capacity of Elderly Women With Knee Osteoarthritis. This is a randomized controlled trial with three allocation groups: spiritual laying on of hands ("passe espiríta" - Spiritist passe/spiritual healing) (SP), non-spiritual laying on of hands (LH) and Control Group without laying on of hands (CG). All subjects will participate in a 45-minute kinesiotherapy program. After that, groups will be directed to the 5-minute session of laying on of hands according to their groups. During the application of SP, LH and CG, the subjects will remain in a sitting position, blindfolded with dark goggles, and receive the following verbal command: "Relax and calm your mind." The intervention will happen twice a week for eight weeks and a blinded physical therapist will assess the pre and post scores of pain, functionality, joint stiffness (through WOMAC and visual analogic scale), anxiety and depression (HADS), religiosity (DUREL) and spirituality (FACIT Sp12) and quality of life (WHOQOL-Bref), among other secondary outcomes.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of chronic degenerative joint disease, as well as the main cause of pain and disability in older persons worldwide. The limited results of the medical and physical therapy approach in the OA treatment make patients with such disorder into possible candidates for complementary and alternative therapies (CAT) aiming to obtain a relieve in their symptoms. Given the importance of providing alternative scientific evidence-based, painless and low cost treatments, it is necessary to carry out studies in order to investigate the impact of CAT in culturally accepted contexts, such as laying on of hands with spiritual or non-spiritual contexts. The present study aims to investigate the effect of Laying on of Hands on the Pain, Joint Stiffness and Functional Capacity of Elderly Women With Knee Osteoarthritis. This is a randomized controlled trial with three allocation groups: spiritual laying on of hands ("passe espiríta" - Spiritist passe/spiritual healing) (SP), non-spiritual laying on of hands (LH) and Control Group without laying on of hands (CG). All subjects will participate in a 45-minute kinesiotherapy program. After that, groups will be directed to the 5-minute session of laying on of hands according to their groups. During the application of SP, LH and CG, the subjects will remain in a sitting position, blindfolded with dark goggles, and receive the following verbal command: "Relax and calm your mind." The intervention will happen twice a week for eight weeks and a blinded physical therapist will assess the pre and post scores of pain, functionality, joint stiffness (through WOMAC and visual analogic scale), anxiety and depression (HADS), religiosity (DUREL) and spirituality (FACIT Sp12) and quality of life (WHOQOL-Bref), among other secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and radiographically diagnosed with OA in both knees, according to the criteria set by the American College of Rheumatology
* Knee OA grade II or III, according to the criteria by Kellgren and Lawrence
* Moderate to very severe pain, according to the Western Ontario and McMaster Universities (WOMAC) pain subscale) (score between 10 and 20)
* Using stable doses of analgesics and NSAIDs during the intervention;
* Do not perform physical therapy or other complementary therapies with laying on of hands different from those proposed in the current study;
* Being able to travel to the rehabilitation site;
* Being able to read, understand and speak Portuguese;
* Preserved cognition

Exclusion Criteria:

* Having made use of oral or intra-articular corticosteroids for at least 3 months before the intervention;
* Having made use of intra-articular hyaluronate for at least three months before the intervention;
* Having full or partial prosthetic hips and/or knees;
* Presenting neurological diseases or other rheumatic diseases;
* Presenting medical contraindications to perform light to moderate physical activity;
* Being absent for two consecutive or three non-consecutive times.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-04 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain on the WOMAC scale | At the beginning, after 8 weeks (end of intervention) and after 16 weeks.
Change from baseline in joint stiffness on the WOMAC scale | At the beginning, after 8 weeks (end of intervention) and after 16 weeks.
Change from baseline in functional capacity on the WOMAC scale | At the beginning, after 8 weeks (end of intervention) and after 16 weeks.
Change from baseline in pain on the visual analog scale | At the beginning, after 8 weeks (end of intervention) and after 16 weeks.

SECONDARY OUTCOMES:
Changes in depressive and anxiety symptoms on the HADS scale | At the beginning, after 8 weeks (end of intervention) and after 16 weeks.
Changes in Quality of life on the WHOQOL-Bref scale | At the beginning, after 8 weeks (end of intervention) and after 16 weeks.
Change from baseline in spirituality on the FACIT Sp12 | At the beginning, after 8 weeks (end of intervention) and after 16 weeks.
Change from baseline in mobility through the "Timed Up and Go" test | At the beginning, after 8 weeks (end of intervention) and after 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Katy A Zacaron, MSc, Principal Investigator — Federal University of Juiz de Fora
Locations (1):
- Juiz de Fora Department of elderly affairs, Juiz de Fora, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zacaron KAM, da Silva Mendes N, E Silva YC, Lucchetti G. Effects of laying on of hands with and without a spiritual context on pain and functionality of older women with knee osteoarthritis: study protocol for a randomized controlled trial. J Integr Med. 2018 Mar;16(2):106-112. doi: 10.1016/j.joim.2018.02.002. Epub 2018 Feb 3. PMID 29526233